CLINICAL TRIAL: NCT05494021
Title: Lung Cancer Screening With Low-dose CT in China (CLUS Study) Version 3.0
Brief Title: China Lung Cancer Screening (CLUS) Study Version 3.0
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Baohui Han, Director, Shanghai Chest Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CLUS 3.0
Record Dates: First submitted 2022-08-07; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole-process management strategy (Experimental): High-risk individuls are provided with whole-process management strategy, including lung cancer education, decision-making, assisting in making and attending LCS LDCT appointments, arranging follow-up when needed, tobacco cessation support for smokers, treatment assistance if diagnosed as lung cancer.
  LDCT was performed at baseline + 2 biennial repeated LDCT rounds.
  Interventions: Other: Whole-process management software; Device: LDCT detection
- Rountine screening strategy (Active Comparator): LDCT was performed at baseline + 2 biennial repeated LDCT rounds.
  Interventions: Device: LDCT detection

INTERVENTIONS:
Other: Whole-process management software — Enrolled participants will managed by a pre-designed software. The software would provide helpful assistance, such as lung cancer education, decision-making, assisting in making and attending LCS LDCT appointments, arranging follow-up when needed, tobacco cessation support for smokers, treatment assistance if diagnosed as lung cancer.
  Arms: Whole-process management strategy
Device: LDCT detection — LDCT were performed in both arm. The abnormal nodules were defined as noncalcified nodules (NCN) larger than 5 mm

SUMMARY:
CLUS version 1.0, had proven that LDCT led to a 74.1% increase in detecting early-stage lung cancer compare to usual care (NCT02898441). CLUS version 2.0 evaluated the efficacy of new techniques (AI, AFI and MTB) in fostering the implementation of lung cancer screening (NCT03975504). The present multi-center study is performed to evaluate the effectiveness of different lung cancer screening strategy and validate our previous findings. 100,000 high-risk subjects (age 45-75) were recruited to take LDCT screening (Baseline + 2 biennial repeated LDCT screening). Follow-up for lung cancer incidence, lung cancer mortality and overall mortality was performed. Blood samples were stored in a Biobank. Management of positive screening test was carried out by a pre-specified protocol.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants were those aged 45-75 years, and with either of the following risk factors:

  1. history of cigarette smoking ≥ 20 pack-years, and, if former smokers, had quit within the previous 15 years;
  2. malignant tumors history in immediate family members;
  3. personal cancer history;
  4. professional exposure to carcinogens;
  5. long term exposure to second-hand smoke;
  6. long term exposure to cooking oil fumes.

Exclusion Criteria:

* Had a CT scan of chest within last 12 months
* History of any cancer within 5 years

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The mortality rate of lung cancer | 5 years
  Assess lung cancer mortality within next 5 years after first round of screening
The attendance rate of high-risk individuals | 5 years
  Evaluate the ability of whole-process management strategy in enhancing the attendance rate of high-risk individuals
The adherence rate of high-risk individuals | 5 years
  Evaluate the ability of whole-process management strategy in enhancing the adherence rate of high-risk individuals

SECONDARY OUTCOMES:
The mortality of all-cause | 5 years
  Assess all-cause mortality within next 5 years after first round of screening
The detection rate of lung nodules | 5 years
  Assess lung nodules detection rate, and the types and sizes of nodules detected in LDCT screening
The incidence rate lung cancer | 5 years
  Assess the number of lung cancer incidences after each round of screening

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No